CLINICAL TRIAL: NCT02844062
Title: A Safety and Efficacy Study of Autologous Chimeric Antigen Receptor Engineered T Cells Redirected to EGFRvIII in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Pilot Study of Autologous Anti-EGFRvIII CAR T Cells in Recurrent Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Sanbo Brain Hospital (Other)
Collaborators: Marino Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBNK-2016-015-01
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-EGFRvIII CAR T cells (Experimental): Patients will receive lymphodepletion chemotherapy consisting of fludarabine and cyclophosphamide, followed by intravenous infusion of autologous anti-EGFRvIII CAR T cells. A standard 3+3 escalation approach will be used to obtain the safe dosage of CAR T cells. The tested CAR T cell dosage ranges from 5×10^4 /kg to 1×10^7 /kg
  Interventions: Biological: anti-EGFRvIII CAR T cells; Drug: cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: anti-EGFRvIII CAR T cells — CAR T cells are infused intravenously to patients in a three-day split-dose regimen（day0,10%; day1, 30%; day2, 60%）with a total targeted dose.
Drug: cyclophosphamide — 250 mg/m^2 d1-3
Drug: Fludarabine — 25mg/m^2 d1-3

SUMMARY:
Chimeric antigen receptor (CAR)-modified T cells can mediate long-term durable remissions in recurrent or refractory CD19+ B cell malignancies, and are a promising therapy to treat glioblastoma, which is the most dangerous and aggressive form of brain cancer. EGFRvIII mutation (epidermal growth factor receptor variant III, EGFRvIII) is the results of tumor specific gene rearrangement naturally happened in about 30% of glioblastoma patients and produces a mutated protein with neo-antigen that is tumor specific and is not expressed in normal human tissues. Therefore, EGFRvIII is an attractive target for CAR T cell therapy. We have constructed a lentiviral vector that contains a chimeric antigen receptor that recognizes the EGFRvIII tumor antigen. A truncated EGFR (tEGFR) which lacks of the ligand binding domain and cytoplasmic kinase domain of wildtype EGFR is incorporated into the CAR vector and is used for in vivo tracking and ablation of CAR T cells in necessary. This pilot study is to determine the safety and efficacy of autologous anti-EGFRvIII CAR T cells in patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. abilities to understand and the willingness to provide written informed consent;
2. patients are ≥ 18 and ≤ 70 years old;
3. recurrent glioblastoma patients with measurable tumors. Patients have received standard care of medication, such as Gross Total Resection with concurrent Radio-chemotherapy (~54 - 60 Gy, TMZ). Patients must either not be receiving dexamethasone or receiving ≤ 4 mg/day at the time of leukopheresis;
4. Malignant cells are EGFRvIII positive confirmed by IHC, quantitative PCR or sequencing;
5. karnofsky performance score (KPS) ≥ 60;
6. life expectancy >3 months;
7. satisfactory bone marrow, liver and kidney functions as defined by the following: absolute neutrophile count ≥ 1500/mm^3; hemoglobin > 10 g/dL; platelets > 100000 /mm^3; Bilirubin < 1.5×ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5×ULN; creatinine < 1.5×ULN;
8. peripheral blood absolute lymphocyte count must be above 0.8×10^9/L;
9. satisfactory heart functions;
10. patients must be willing to follow the orders of doctors;
11. women of reproductive potential (between 15 and 49 years old) must have a negative pregnancy test within 7 days of study start. Male and female patients of reproductive potential must agree to use birth control during the study and 3 months post study.

Exclusion Criteria:

1. a prior history of gliadel implantation 4 weeks before this study start or antibody based therapies;
2. HIV positive;
3. hepatitis B infection or hepatitis C infection;
4. history of autoimmune disease, or other diseases require long-term administration of steroids or immunosuppressive therapies;
5. history of allergic disease, or allergy to CAR T cells or study product excipients;
6. patients already enrolled in other clinical study;
7. patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion of autologous anti-EGFRvIII CAR T cells with cyclophosphamide and fludarabine as lymphodepleting chemotherapy in patients with recurrent glioblastoma using the NCI CTCAE V4.0 criteria. | 2 years
  incidents of treatment related adverse events as assessed by CTCAE V4.0.

SECONDARY OUTCOMES:
Treatment Responses Rate | 4 weeks
  defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD).
Overall Survival Rate | 2 years
Progression-free Survival Rate | 2 years
Persistence of CAR T cells in patients | 2 years

OTHER OUTCOMES:
Proliferation of CAR T cells in patients | 2 years
  CAR T cell proliferation in patients is monitored by flow or qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiong Lin, MD, Principal Investigator — Capital Medical University
Locations (1):
- Sanbo Brain Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes